CLINICAL TRIAL: NCT02061761
Title: A Phase 1/2a Dose Escalation and Cohort Expansion Study of the Safety, Tolerability, and Efficacy of Anti-LAG-3 Monoclonal Antibody (Relatlimab, BMS-986016) Administered Alone and in Combination With Anti-PD-1 Monoclonal Antibody (Nivolumab, BMS-936558) in Relapsed or Refractory B-Cell Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of Relatlimab in Relapsed or Refractory B-Cell Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA224-022
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Hematologic Neoplasms
Keywords: Hodgkin lymphoma; non-Hodgkin lymphoma; diffused large B-cell lymphoma; indolent lymphoma; chronic lymphocytic leukemia; relapsed; refractory
MeSH Terms: conditions — Hematologic Neoplasms; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A - relatlimab (Dose escalation) (Experimental)
  Interventions: Biological: BMS-986016
- Part C - relatlimab + nivolumab (Dose escalation) (Experimental)
  Interventions: Biological: BMS-986016; Biological: BMS-936558
- Part B - relatlimab (Cohort expansion) (Experimental)
  Interventions: Biological: BMS-986016
- Part D - relatlimab + nivolumab (Cohort expansion) (Experimental)
  Interventions: Biological: BMS-986016; Biological: BMS-936558

INTERVENTIONS:
Biological: BMS-986016 — Specified Dose on Specified Days
  Other Names: Anti-LAG-3 (Anti-Lymphocyte Activation Gene-3), relatlimab
Biological: BMS-936558 — Specified Dose on Specified Days
  Other Names: Anti-PD-1 (Anti-Programmed-Death-1), MDX-1106, nivolumab
  Arms: Part C - relatlimab + nivolumab (Dose escalation); Part D - relatlimab + nivolumab (Cohort expansion)

SUMMARY:
The primary objective of this study is to characterize the safety, tolerability, dose-limiting toxicities (DLTs), and maximum tolerated dose (MTD) of relatlimab administered alone or in combination with nivolumab to subjects with relapsed or refractory B-cell malignancies. Co-primary objective is to investigate the preliminary efficacy of relatlimab in combination with nivolumab in subjects with relapsed or refractory Hodgkin lymphoma (HL), and relapsed or refractory Diffused Large B Cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Must have histologic or cytologic confirmation of chronic lymphocytic leukemia, Hodgkin lymphoma, Non-Hodgkin lymphoma, or Multiple Myeloma and have relapsed following prior treatment or been refractory to prior treatment
* Must have progressed or been refractory to, at least one prior standard therapy, including radiation, immunomodulatory agents (eg, lenalidomide), immunotherapy, cytotoxic chemotherapy, and select antibody (anti-CD20, alemtuzumab, or anti-CD30) therapy.
* Must be more than 100 days post autologous transplant

Exclusion Criteria:

* Known or suspected central nervous system (CNS) metastases or with the CNS as the only site of active disease (controlled CNS metastases are allowed)
* Known or suspected autoimmune disease
* History of allergy to anti-PD-1 or anti-PD-L1 antibody therapy or to other monoclonal antibodies or related compounds or to any of their components

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (8):
  - Local Institution - 0007, Baltimore, Maryland
  - Local Institution - 0004, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Local Institution - 0010, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Local Institution - 0002, Portland, Oregon
  - Local Institution - 0006, Houston, Texas
  - Local Institution - 0001, Seattle, Washington
- Canada (2):
  - Local Institution - 0011, Vancouver, British Columbia
  - Local Institution - 0012, Toronto, Ontario

REFERENCES:
- [Derived] Gopal AK, Armand P, Neelapu SS, Bartlett NL, Spurgeon SE, Kuruvilla J, Savage KJ, Leonard JP, Gelb AB, Ahmed N, Dong S, Bathena SP, Suryawanshi R, Wu JQ, Wang S, Gladstone DE. Nivolumab plus relatlimab for patients with relapsed or progressed B-cell malignancies in RELATIVITY-022. Blood Adv. 2025 Jul 8;9(13):3383-3394. doi: 10.1182/bloodadvances.2024015086. PMID 40030000
- [Derived] El Halabi L, Adam J, Gravelle P, Marty V, Danu A, Lazarovici J, Ribrag V, Bosq J, Camara-Clayette V, Laurent C, Ghez D. Expression of the Immune Checkpoint Regulators LAG-3 and TIM-3 in Classical Hodgkin Lymphoma. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):257-266.e3. doi: 10.1016/j.clml.2020.11.009. Epub 2020 Nov 12. PMID 33277223
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986016 20mg: Dose escalation (part A): BMS-986016 20mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 80mg: Dose escalation (part A): BMS-986016 80mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 800mg: Dose escalation (part A): BMS-986016 800mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 240mg: Dose escalation (part A): BMS-986016 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 240mg Part B: Dose expansion (part B): BMS-986016 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 80mg + Nivolumab: Dose escalation (part C): BMS-986016 IV 80mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 240mg + Nivolumab: Dose escalation (part C): BMS-986016 IV 240mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 160mg + Nivolumab: Dose escalation (part C): BMS-986016 IV 160mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 160mg + Nivolumab Part D: Dose expansion (part D): BMS-986016 IV 160mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
Period: Overall Study
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 240mg Part B | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab | BMS-986016 160mg + Nivolumab Part D
Started (Started treatment) | 3 | 9 | 6 | 9 | 11 | 7 | 1 | 4 | 56
Chronic Lymphocytic Leukemia (CLL) (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Diffuse Large B-Cell Lymphoma (DLBCL) (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 15
Indolent Non-Hodgkin Lymphoma (iNHL) (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Hodgkin Lymphoma (HL) (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
HL-anti-PD-1 Naive (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
HL-anti-PD-1 Progressed (Tumor type eligible for expansion) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Completed (Completed treatment) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 5
Not Completed | 3 | 8 | 6 | 9 | 11 | 5 | 1 | 4 | 51
Not completed — Disease progression | 2 | 8 | 4 | 5 | 9 | 3 | 1 | 2 | 28
Not completed — Study Drug toxicity | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 6
Not completed — Adverse event unrelated to study Drug | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant request to discontinue study treatment | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Maximum clinical benefit | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6
Not completed — Participant no longer meets study criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other reasons | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- BMS-986016 240mg: Dose escalation (part A) and dose expansion (part B): BMS-986016 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- BMS-986016 160mg + Nivolumab: Dose escalation (part C) and dose expansion (part D): BMS-986016 IV 160mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, until meeting criteria for discontinuation, or clinical deterioration, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- Total: Total of all reporting groups
Arm/Group | BMS-986016 20mg | BMS-986016 800mg | BMS-986016 80mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab | Total
Number analyzed (Participants) | 3 | 9 | 6 | 20 | 7 | 1 | 60 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5 | 12 | 3 | 1 | 46 | 72
  >=65 years | 1 | 6 | 1 | 8 | 4 | 0 | 14 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 1 | 6 | 4 | 0 | 22 | 38
  Male | 3 | 4 | 5 | 14 | 3 | 1 | 38 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Not Hispanic or Latino | 3 | 9 | 5 | 19 | 7 | 1 | 58 | 102
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 1 | 2 | 0 | 0 | 4 | 9
  White | 1 | 8 | 5 | 16 | 7 | 1 | 45 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 0 | 0 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: Number of participants with any grade adverse events (AEs), any grade serious adverse events (SAEs) and any grade AEs leading to discontinuation of any drug. The severity of AEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 100 days post last dose (Up to 51 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 9 | 6 | 20 | 7 | 1 | 60
Participants
  AEs | 3 | 9 | 5 | 19 | 7 | 1 | 59
  SAEs | 1 | 4 | 2 | 6 | 4 | 0 | 26
  AEs leading to discontinuation | 1 | 2 | 0 | 1 | 1 | 0 | 9

2. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: From first dose to 135 days post last dose (Up to 52 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 9 | 6 | 20 | 7 | 1 | 60
Participants | 0 | 2 | 1 | 2 | 2 | 0 | 10

3. Primary Outcome: Number of Participants With On-Treatment Laboratory Abnormalities in Specific Hepatics Tests
Description: Number of participants with laboratory abnormalities in specific hepatic tests based on SI unit convention. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * ALP > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to 30 days post last dose (Up to 49 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 9 | 5 | 20 | 7 | 1 | 57
Participants
  ALT OR AST > 3XULN | 0 | 0 | 0 | 0 | 0 | 0 | 5
  ALT OR AST > 5XULN | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT OR AST > 10XULN | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT OR AST > 20XULN | 0 | 0 | 0 | 0 | 0 | 0 | 1
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 0 | 1 | 0 | 0 | 1
  ALP > 1.5XULN | 1 | 1 | 0 | 1 | 1 | 0 | 8
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN ONE DAY | 0 | 0 | 0 | 0 | 0 | 0 | 2
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 1.5XULN WITHIN 30 DAYS | 0 | 0 | 0 | 0 | 0 | 0 | 2
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN ONE DAY | 0 | 0 | 0 | 0 | 0 | 0 | 1
  CONCURRENT ALT OR AST ELEVATION > 3XULN WITH TOTAL BILIRUBIN > 2XULN WITHIN 30 DAYS | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Objective Response Rate (ORR) - Part D
Description: Investigator-assessed ORR per International Working Group (IWG 2007) response criteria for malignant lymphoma is defined as the number of participants with a best overall documented response (BOR) of either a complete response (CR) or partial response (PR).
  Complete response: Disappearance of all evidence of disease. Partial response: Regression of measurable disease and no new sites. >= 50% decrease in sum of the produce of the diameters of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions).
  Progressive disease: Any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: From first dose date to the date of disease progression per investigator or the date of subsequent therapy, whichever occurs first (Up to approximately 95 months)
Population: Pre-specified only to be collected in all treated participants by tumor type for Part D
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HL Naive BMS-986016 160mg + Nivolumab; DLBCL BMS-986016 160mg + Nivolumab; HL Post I/O BMS-986016 160mg + Nivolumab: Dose expansion (part D): BMS-986016 IV 160mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
Arm/Group | HL Naive BMS-986016 160mg + Nivolumab | DLBCL BMS-986016 160mg + Nivolumab | HL Post I/O BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 21 | 15 | 20
Percentage of participants | 61.9 [38.4 to 81.9] | 6.7 [0.2 to 31.9] | 15.0 [3.2 to 37.9]

5. Primary Outcome: Duration of Response (DoR) - Part D
Description: Investigator-assessed DoR per International Working Group (IWG 2007)) response criteria for malignant lymphoma is defined as the time between the date of first documented response (complete response or partial response) to the date of the first objectively documented progression, or death due to any cause, whichever occurs first.
  Complete response: Disappearance of all evidence of disease. Partial response: Regression of measurable disease and no new sites. >= 50% decrease in sum of the produce of the diameters of up to 6 largest dominant masses (index lesions); no increase in size of other nodes (non-index lesions).
  Progressive disease: Any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: From first dose to the date of the first objectively documented progression, or death due to any cause, whichever occurs first (Up to approximately 95 months)
Population: Pre-specified only to be collected in all responders (CR or PR) by tumor type for Part D
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HL Naive BMS-986016 160mg + Nivolumab | DLBCL BMS-986016 160mg + Nivolumab | HL Post I/O BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 13 | 1 | 3
Months | 14.16 [2.56 to NA] — Upper limit not available due to insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events | 6.37 [1.84 to NA] — Upper limit not available due to insufficient number of participants with events

6. Secondary Outcome: BMS-986016 Maximum Observed Serum Concentration (Cmax)
Description: BMS-986016 Maximum Observed Serum Concentration (Cmax). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: PK assessment include the following timepoints: pre-dose, 1, 4, 24, 48, 96, 144, 192 hours end-of-infusion on cycle 1 Day 1, Cycle 3 Day 1
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 6 | 20 | 7 | 1 | 37
ug/mL
  Period 0, Cycle 1, Day 1 (P0C1D1) | 3.697 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40 | 22.738 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 29 | 224.802 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 32 | 68.718 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 54 | 19.990 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 25 | 57.900 (NA) — insufficient numbers of participants with events | 40.402 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26
  P0C3D1: number analyzed (Participants) | 2 | 2 | 1 | 7 | 3 | 1 | 13
  P0C3D1 | 6.660 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 21 | 31.917 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 81 | 673.000 (NA) — insufficient numbers of participants with events | 116.419 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 49 | 44.532 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 12 | 149.000 (NA) — insufficient numbers of participants with events | 88.196 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 44
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D1 |  |  |  |  |  | 59.600 (NA) — insufficient numbers of participants with events | 68.400 (NA) — insufficient numbers of participants with events
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 165.000 (NA) — insufficient numbers of participants with events | 163.000 (NA) — insufficient numbers of participants with events

7. Secondary Outcome: BMS-986016 Time of Maximum Observed Serum Concentration (Tmax)
Description: BMS-986016 Time of Maximum Observed Serum Concentration (Tmax). Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 6 | 20 | 7 | 1 | 37
Hours
  Period 0, Cycle 1, Day 1 (P0C1D1) | 0.97 [0.97 to 0.97] | 1.300 [1.00 to 4.00] | 4.167 [1.00 to 24.00] | 1.825 [0.97 to 95.75] | 3.950 [1.00 to 5.00] | 0.97 [0.97 to 0.97] | 1.600 [0.97 to 24.07]
  P0C3D1: number analyzed (Participants) | 2 | 2 | 1 | 7 | 3 | 1 | 13
  P0C3D1 | 0.984 [0.97 to 1.00] | 10.975 [1.37 to 20.58] | 168.22 [168.22 to 168.22] | 1.233 [0.97 to 23.87] | 1.017 [1.00 to 4.00] | 1.000 [1.00 to 1.00] | 3.467 [0.92 to 46.45]
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D1 |  |  |  |  |  | 4.000 [4.00 to 4.00] | 1.750 [1.75 to 1.75]
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 24.000 [24.00 to 24.00] | 0.900 [0.90 to 0.90]

8. Secondary Outcome: BMS-986016 Area Under the Concentration-time Curve in One Dosing Interval (AUC(TAU))
Description: BMS-986016 Area under the concentration-time curve in one dosing interval (AUC(TAU)). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 6 | 20 | 7 | 1 | 37
h*ug/mL
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 3 | 7 | 5 | 18 | 7 | 1 | 26
  Period 0, Cycle 1, Day 1 (P0C1D1) | 401.438 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 38 | 2852.533 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57 | 44296.525 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 20 | 9086.827 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 41 | 2908.011 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 38 | 9480.758 (NA) — insufficient numbers of participants with events | 5327.954 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40
  P0C3D1: number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
  P0C3D1 | 712.408 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 6 | 4898.034 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 116 | 176405.369 (NA) — insufficient numbers of participants with events | 18783.970 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 87 | 6166.165 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 64 | 34573.957 (NA) — insufficient numbers of participants with events | 20464.075 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 48
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D1 |  |  |  |  |  | 11259.871 (NA) — insufficient numbers of participants with events | 11433.253 (NA) — insufficient numbers of participants with events
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 38472.003 (NA) — insufficient numbers of participants with events | 33919.259 (NA) — insufficient numbers of participants with events

9. Secondary Outcome: BMS-986016 Concentration at the End of a Dosing Interval (Ctau)
Description: BMS-986016 Concentration at the end of a dosing interval (Ctau). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 5 | 18 | 7 | 1 | 26
h*ug/mL
  Period 0, Cycle 1, Day 1 (P0C1D1) | 0.158 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 79 | 1.037 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 86 | 75.589 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31 | 12.221 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 75 | 3.848 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 53 | 19.500 (NA) — insufficient numbers of participants with events | 8.417 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57
  P0C3D1: number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
  P0C3D1 | 0.256 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 125 | 2.266 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 140 | 293.000 (NA) — insufficient numbers of participants with events | 30.970 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 110 | 9.556 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 78 | 103.000 (NA) — insufficient numbers of participants with events | 47.016 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 54
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D1 |  |  |  |  |  | 25.900 (NA) — insufficient numbers of participants with events | 24.200 (NA) — insufficient numbers of participants with events
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 86.600 (NA) — insufficient numbers of participants with events | 86.100 (NA) — insufficient numbers of participants with events

10. Secondary Outcome: BMS-986016 Effective Elimination Half-life That Explains the Degree of AUC Accumulation Observed (T 1/2eff AUC)
Description: BMS-986016 effective elimination half-life that explains the degree of AUC accumulation observed (t 1/2eff AUC). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 1 | 1 | 5 | 2 | 1 | 12
Hours
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 240.671 (143.5338) | 742.843 (NA) — insufficient numbers of participants with events | 547.986 (NA) — insufficient numbers of participants with events | 428.698 (346.4046) | 548.741 (78.0213) | 720.317 (NA) — insufficient numbers of participants with events | 674.755 (296.9473)
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 638.597 (NA) — insufficient numbers of participants with events | 524.637 (NA) — insufficient numbers of participants with events

11. Secondary Outcome: BMS-986016 Total Body Clearance (CL/T)
Description: BMS-986016 total body clearance (CL/T). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 = Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
mL/h
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 28.074 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 6 | 16.333 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 116 | 4.535 (NA) — insufficient numbers of participants with events | 12.777 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 75 | 12.974 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 96 | 6.942 (NA) — insufficient numbers of participants with events | 7.819 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 41
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 6.238 (NA) — insufficient numbers of participants with events | 4.717 (NA) — insufficient numbers of participants with events

12. Secondary Outcome: BMS-986016 Cmax Accumulation Index (AI_Cmax)
Description: BMS-986016 cmax accumulation index (AI_Cmax). AI is calculated based on ratio of Cmax at steady state to Cmax after the first dose. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 - Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 2 | 1 | 7 | 3 | 1 | 12
ug/mL
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 1.981 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40 | 1.701 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 68 | 2.009 (NA) — insufficient numbers of participants with events | 1.734 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 42 | 2.369 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 12 | 2.573 (NA) — insufficient numbers of participants with events | 2.139 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 28
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 2.768 (NA) — insufficient numbers of participants with events | 2.383 (NA) — insufficient numbers of participants with events

13. Secondary Outcome: BMS-986016 Accumulation Index (AI_AUC)
Description: BMS-986016 accumulation index (AI_AUC). AI is calculated based on ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 - Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
Ratio
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 1.577 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 34 | 1.850 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 86 | 2.894 (NA) — insufficient numbers of participants with events | 2.186 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 58 | 2.017 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 50 | 3.647 (NA) — insufficient numbers of participants with events | 3.268 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 32
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 3.417 (NA) — insufficient numbers of participants with events | 2.967 (NA) — insufficient numbers of participants with events

14. Secondary Outcome: BMS-986016 Ctau Accumulation Index (AI_Ctau)
Description: BMS-986016 Ctau accumulation index (AI_Ctau). AI is calculated based on ratio of Ctau at steady state to Ctau after the first dose. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 - Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
Ratio
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 0.743 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =118 | 2.494 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 74 | 4.741 (NA) — insufficient numbers of participants with events | 2.310 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 68 | 1.686 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 69 | 5.282 (NA) — insufficient numbers of participants with events | 4.162 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 26
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 3.344 (NA) — insufficient numbers of participants with events | 3.558 (NA) — insufficient numbers of participants with events

15. Secondary Outcome: BMS-986016 Average Concentration Over a Dosing Interval ([AUC(TAU)/Tau] (Css,Avg)
Description: BMS-986016 average concentration over a dosing interval ([AUC(TAU)/tau] (Css,avg). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 - Re-challenge period
Time Frame: as for outcome 6
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 2 | 2 | 1 | 5 | 3 | 1 | 12
ug/mL
  Period 0, Cycle 1, Day 1 (P0C1D1): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P0C3D1 | 2.117 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =6 | 14.738 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 116 | 526.269 (NA) — insufficient numbers of participants with events | 57.790 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 85 | 18.345 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 64 | 103.805 (NA) — insufficient numbers of participants with events | 61.385 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 46
  P1C1D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 120.595 (NA) — insufficient numbers of participants with events | 109.013 (NA) — insufficient numbers of participants with events

16. Secondary Outcome: BMS-986016 Trough Observed Serum Concentration (Ctrough)
Description: BMS-986016 trough observed serum concentration (Ctrough). Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
  Period 0 = treatment period Period 1 - Re-challenge period
Time Frame: PK assessment include the following timepoints: pre-dose, 1, 4, 24, 48, 96, 144, 192 hours end-of-infusion on cycle 1 Day 15, 29, 43, Cycle 2 Day 1, 15, 29, Cycle 3 Day 1, 15, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1, and Cycle 11 Day 1
Population: All participants who received at least one dose of BMS-986016 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 5 | 19 | 7 | 1 | 48
ug/mL
  P0C1D15: number analyzed (Participants) | 3 | 7 | 5 | 18 | 7 | 1 | 44
  P0C1D15 | 0.064 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =145 | 1.457 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 85 | 75.589 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 31 | 12.221 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 75 | 3.848 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 53 | 19.500 (NA) — insufficient numbers of participants with events | 10.609 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 46
  P0C1D29: number analyzed (Participants) | 3 | 6 | 5 | 19 | 4 | 1 | 48
  P0C1D29 | 0.088 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =141 | 4.324 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =78 | 155.896 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 33 | 20.982 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 78 | 13.066 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 17 | 32.400 (NA) — insufficient numbers of participants with events | 18.221 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 41
  P0C1D43: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 1 | 37
  P0C1D43 |  |  |  |  | 9.435 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 55 | 44.700 (NA) — insufficient numbers of participants with events | 25.234 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43
  P0C2D1: number analyzed (Participants) | 2 | 4 | 4 | 14 | 3 | 1 | 34
  P0C2D1 | 0.777 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =141 | 6.609 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =75 | 298.666 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43 | 37.013 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 114 | 9.389 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 74 | 59.000 (NA) — insufficient numbers of participants with events | 28.428 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43
  P0C2D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1 | 25
  P0C2D15 |  |  |  |  | 6.209 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 123 | 62.000 (NA) — insufficient numbers of participants with events | 30.218 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 45
  P0C2D29: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 1 | 6
  P0C2D29 |  |  | 289.000 (NA) — insufficient numbers of participants with events |  | 26.700 (NA) — insufficient numbers of participants with events | 70.900 (NA) — insufficient numbers of participants with events | 36.675 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 50
  P0C3D1: number analyzed (Participants) | 1 | 2 | 1 | 7 | 2 | 1 | 21
  P0C3D1 | 1.020 (NA) — insufficient numbers of participants with events | 19.018 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =86 | 313.000 (NA) — insufficient numbers of participants with events | 16.648 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 121 | 6.867 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 125 | 93.300 (NA) — insufficient numbers of participants with events | 45.535 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 46
  P0C3D15: number analyzed (Participants) | 2 | 2 | 1 | 6 | 3 | 1 | 23
  P0C3D15 | 0.256 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =125 | 2.266 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =140 | 293.000 (NA) — insufficient numbers of participants with events | 9.450 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 127 | 9.556 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 78 | 103.000 (NA) — insufficient numbers of participants with events | 45.685 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 48
  P0C5D1: number analyzed (Participants) | 2 | 2 | 0 | 3 | 2 | 1 | 14
  P0C5D1 | 0.729 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =45 | 1.917 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =141 |  | 18.198 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV =81 | 23.381 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 41 | 149.000 (NA) — insufficient numbers of participants with events | 57.068 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 56
  P0C7D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 2 | 1 | 6
  P0C7D1 |  | 59.600 (NA) — insufficient numbers of participants with events |  | 5.760 (NA) — insufficient numbers of participants with events | 20.264 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 70 | 143.000 (NA) — insufficient numbers of participants with events | 58.408 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40
  P0C9D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 1 | 4
  P0C9D1 |  | 62.000 (NA) — insufficient numbers of participants with events |  | 5.860 (NA) — insufficient numbers of participants with events | 22.800 (NA) — insufficient numbers of participants with events | 117.000 (NA) — insufficient numbers of participants with events | 56.054 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 62
  P0C11D1: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 1 | 3
  P0C11D1 |  | 48.100 (NA) — insufficient numbers of participants with events |  | 4.710 (NA) — insufficient numbers of participants with events | 31.200 (NA) — insufficient numbers of participants with events | 165.000 (NA) — insufficient numbers of participants with events | 67.268 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 64
  P1C1D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D15 |  |  |  |  |  | 25.900 (NA) — insufficient numbers of participants with events | 24.200 (NA) — insufficient numbers of participants with events
  P1C1D29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D29 |  |  |  |  |  | 43.600 (NA) — insufficient numbers of participants with events | 41.000 (NA) — insufficient numbers of participants with events
  P1C1D43: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C1D43 |  |  |  |  |  | 61.800 (NA) — insufficient numbers of participants with events | 56.000 (NA) — insufficient numbers of participants with events
  P1C2D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C2D1 |  |  |  |  |  | 73.800 (NA) — insufficient numbers of participants with events | 58.700 (NA) — insufficient numbers of participants with events
  P1C2D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C2D15 |  |  |  |  |  | 84.700 (NA) — insufficient numbers of participants with events | 69.400 (NA) — insufficient numbers of participants with events
  P1C2D29: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C2D29 |  |  |  |  |  | 81.500 (NA) — insufficient numbers of participants with events | 71.900 (NA) — insufficient numbers of participants with events
  P1C3D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D1 |  |  |  |  |  | 94.600 (NA) — insufficient numbers of participants with events | 85.500 (NA) — insufficient numbers of participants with events
  P1C3D15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C3D15 |  |  |  |  |  | 86.600 (NA) — insufficient numbers of participants with events | 86.100 (NA) — insufficient numbers of participants with events
  P1C5D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C5D1 |  |  |  |  |  | 109.000 (NA) — insufficient numbers of participants with events | 70.100 (NA) — insufficient numbers of participants with events
  P1C7D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C7D1 |  |  |  |  |  | 107.000 (NA) — insufficient numbers of participants with events | 105.000 (NA) — insufficient numbers of participants with events
  P1C9D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 1
  P1C9D1 |  |  |  |  |  | 115.000 (NA) — insufficient numbers of participants with events | 110.000 (NA) — insufficient numbers of participants with events
  P1C11D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  P1C11D1 |  |  |  |  |  |  | 115.000 (NA) — insufficient numbers of participants with events

17. Secondary Outcome: Number of Participants With Anti-BMS-986016 Antibodies (ADA)
Description: Number of participants with anti-BMS-986016 antibodies (ADA) with status as baseline ADA positive, ADA positive and ADA negative. Baseline ADA positive participant is defined as a participant with positive seroconversion detected in the last sample before initiation of treatment. ADA-positive participant is a participant with at least one ADA-positive sample relative to baseline after initiation of the treatment. ADA negative participant is defined as a participant with no ADA positive sample after the initiation of treatment.
Time Frame: From first dose to 135 days post last dose (Up to 52 months)
Population: All BMS-986016 treated participants with baseline and at least one post-baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 3 | 7 | 5 | 19 | 7 | 1 | 52
Participants
  Baseline ADA Positive | 0 | 1 | 1 | 6 | 0 | 0 | 5
  ADA Positive | 0 | 0 | 0 | 7 | 3 | 0 | 4
  ADA Negative | 3 | 7 | 5 | 12 | 4 | 1 | 48

18. Secondary Outcome: Number of Participants With Anti-Nivolumab Antibodies (ADA)
Description: Number of participants with anti-Nivolumab antibodies (ADA) with status as baseline ADA positive, ADA positive and ADA negative. Baseline ADA positive participant is defined as a participant with positive seroconversion detected in the last sample before initiation of treatment. ADA-positive participant is a participant with at least one ADA-positive sample relative to baseline after initiation of the treatment. ADA negative participant is defined as a participant with no ADA positive sample after the initiation of treatment.
Time Frame: From first dose to 135 days post last dose (Up to 52 months)
Population: All Nivolumab treated participants with baseline and at least one post-baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986016 20mg | BMS-986016 80mg | BMS-986016 800mg | BMS-986016 240mg | BMS-986016 80mg + Nivolumab | BMS-986016 240mg + Nivolumab | BMS-986016 160mg + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 1 | 46
Participants
  Baseline ADA Positive |  |  |  |  | 0 | 0 | 0
  ADA Positive |  |  |  |  | 0 | 0 | 1
  ADA Negative |  |  |  |  | 4 | 1 | 45

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) and Other (Not including Serious) Adverse Events (AEs) are collected from first dose to 135 days post last dose (Up to 52 months). Participants were assessed for All-cause mortality from their date of randomization to study completion (Up to approximately 95 months).
Groups:
- All Mono Esc 20 Q2W; All Mono Esc 80 Q2W; All Mono Esc 240 Q2W; All Mono Esc 800 Q2W: Dose escalation (part A): BMS-986016 800mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- CLL BMS-986016 240mg; DLBCL BMS-986016 240mg; iNHL BMS-986016 240mg; HL BMS-986016 240mg: Dose expansion (part B): BMS-986016 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of BMS-986016 administered on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- All Combo Esc 80/240 Q2W: Dose escalation (part C): BMS-986016 IV 80mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- All Combo Esc 160/240 Q2W: Dose escalation (part C): BMS-986016 IV 160mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
- All Combo Esc 240/240 Q2W: Dose escalation (part C): BMS-986016 IV 240mg + Nivolumab IV 240mg up to twelve 8-week treatment cycles, confirmed progressive disease, or until meeting criteria for discontinuation, whichever occurs first. Each treatment cycle comprises 4 doses of Nivolumab followed by BMS-986016 on days 1, 15, 29, and 43. Participants could further receive therapy for up to 6 additional eight-week cycles if re-challenge period criteria are met.
Arm/Group | All Mono Esc 20 Q2W | All Mono Esc 80 Q2W | All Mono Esc 240 Q2W | All Mono Esc 800 Q2W | CLL BMS-986016 240mg | DLBCL BMS-986016 240mg | iNHL BMS-986016 240mg | HL BMS-986016 240mg | All Combo Esc 80/240 Q2W | All Combo Esc 160/240 Q2W | All Combo Esc 240/240 Q2W | HL Naive BMS-986016 160mg + Nivolumab | DLBCL BMS-986016 160mg + Nivolumab | HL Post I/O BMS-986016 160mg + Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/9 | 0/9 | 1/6 | 1/2 | 2/2 | 0/4 | 0/3 | 5/7 | 2/4 | 0/1 | 1/21 | 13/15 | 3/20
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/9 | 1/9 | 2/6 | 1/2 | 2/2 | 2/4 | 1/3 | 4/7 | 2/4 | 0/1 | 6/21 | 11/15 | 9/20
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 8/9 | 5/6 | 2/2 | 2/2 | 4/4 | 3/3 | 7/7 | 4/4 | 1/1 | 20/21 | 11/15 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Mono Esc 20 Q2W (N=3) | All Mono Esc 80 Q2W (N=9) | All Mono Esc 240 Q2W (N=9) | All Mono Esc 800 Q2W (N=6) | CLL BMS-986016 240mg (N=2) | DLBCL BMS-986016 240mg (N=2) | iNHL BMS-986016 240mg (N=4) | HL BMS-986016 240mg (N=3) | All Combo Esc 80/240 Q2W (N=7) | All Combo Esc 160/240 Q2W (N=4) | All Combo Esc 240/240 Q2W (N=1) | HL Naive BMS-986016 160mg + Nivolumab (N=21) | DLBCL BMS-986016 160mg + Nivolumab (N=15) | HL Post I/O BMS-986016 160mg + Nivolumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 1 | 9 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis autoimmune (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Mono Esc 20 Q2W (N=3) | All Mono Esc 80 Q2W (N=9) | All Mono Esc 240 Q2W (N=9) | All Mono Esc 800 Q2W (N=6) | CLL BMS-986016 240mg (N=2) | DLBCL BMS-986016 240mg (N=2) | iNHL BMS-986016 240mg (N=4) | HL BMS-986016 240mg (N=3) | All Combo Esc 80/240 Q2W (N=7) | All Combo Esc 160/240 Q2W (N=4) | All Combo Esc 240/240 Q2W (N=1) | HL Naive BMS-986016 160mg + Nivolumab (N=21) | DLBCL BMS-986016 160mg + Nivolumab (N=15) | HL Post I/O BMS-986016 160mg + Nivolumab (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 4 | 2 | 5
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Eye oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Anal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 3 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 5 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 0 | 4 | 1 | 4
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 5 | 1 | 1
Application site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2
Fatigue (General disorders) | 1 | 4 | 6 | 2 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 8 | 4 | 8
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Oedema peripheral (General disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 4 | 1 | 6
Vaccination site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal foot infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 6 | 1 | 4
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Device placement issue (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 3
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 6 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 3
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 4 | 3 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 5 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 5 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 8 | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lichen planus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 8 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT02061761/Prot_SAP_000.pdf